CLINICAL TRIAL: NCT04918602
Title: Development of Predictive Models Based on Artificial Intelligence for the Analysis of the Psychosocial Profile of the Patient With Fibromyalgia on Pain and Severity of the Disease.
Brief Title: Predictive Models on Pain and Severity in FM Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: IA Fibromyalgia
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this research project is to develop different prediction models in fibromyalgia disease through the application of machine learning techniques and to assess the explainability of the results.

As specific objectives the research project intends: to predicting Fibromyalgia severity of patients based on clinical variables; to assess the relevance of social-psycho-demographic variables on the fibromyalgia severity of the patients; to predict the pain suffered by the patients as well as the impact of the fibromyalgia on patient's life; to categorize fibromyalgia group of patients depending on their levels of Fibromyalgia severity.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a condition characterized by chronic musculoskeletal pain whose pathophysiology is still unclear. Furthermore, this pathology is frequently associated with sleep disturbances, pronounced fatigue, morning stiffness, poor quality of life, cognitive disturbances (mainly memory problems) and psychological problems (depression, anxiety and stress).

FM is associated with greater negative affect, which implies a general state of anguish composed of aversive emotions such as sadness, fear, anger and guilt. Patients with FM commonly suffer from high rates of anxiety, depression, pain catastrophizing, and stress levels, which are associated with a worsening of symptoms, including own cognitive.

Machine learning (ML) and data mining had been successfully applied, over the past few decades, to build computer-aided diagnosis (CAD) systems for diagnosing complex health issues with good accuracy and efﬁciency by recognizing potentially useful, original, and comprehensible patterns in health data. Thus, machine learning provides useful tools for multivariate data analysis allowing predictions based on the established models and hence offering a suitable advantage for risk assessment of many diseases including heart failure. Machine learning offers advantages not only for clinical prediction but also for feature ranking improving the interpretation of the outputs by clinical professionals.

Explainable ML models, also known as interpretable ML models, allow healthcare experts to make reasonable and data-driven decisions to provide personalized treatment that can ultimately lead to high quality of service in healthcare. These models fall into eXplainable Artificial Intelligence (XAI) field, defined as suite of ML techniques that 1) produce more explainable models while maintaining a high level of learning performance, and 2) enable humans to understand, appropriately trust, and eﬀectively manage the emerging generation of artiﬁcially intelligent partners.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Fullfilled the 2010 American Collegue of Rheumathology criteria for fibromyalgia.
* Understanding of spoken and written Spanish.

Exclusion Criteria:

* Diagnosed psychiatric pathology.
* Rheumatic pathology not medically controlled.
* Neurological pathologies that make evaluations difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members enrolled in a local fibromyalgia association.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline.
  It will be measured with a visual analog scale (VAS) of 100 millimeters in length. The subject has to indicate the level ofpain he feels, being 0 the absence of pain and 100 the maximum imaginable.
Disease severity. | Baseline.
  It will be measured using the Polysymptomatic Distress Scale (PDS) (or Fibromyalgia Severity Scale), composed of the sum of the following two scales:
  1. Widespread Pain Index (WPI): Questionnaire in which a total of 19 body areas are represented. The subject has to mark the regions where the pain appears. It represents a measure of the extent of pain, with a maximum score of 19 points.
  2. Symptom Severity Scale (SSS): Questionnaire that measures the severity of the symptoms associated with fibromyalgia, such as fatigue, non-restorative sleep, cognitive problems, headaches, abdominal pain or cramps and depression. It represents a measure of somatic and non-somatic symptoms of fibromyalgia, with a maximum score of 12 points.
Referred pain area after suprathreshold pressure stimulation. | Baseline.
  A pressure algometer (Force Ten™, Wagner Instruments, USA) will be used. It will be performed on the infraspinatus muscle (point equidistant between the midpoint of the spine of the scapula, the inferior angle of the scapula and the midpoint of the medial border of the scapula) at a constant suprathreshold pressure (20% above the pressure pain threshold) for 60 seconds.
  After the stimulation, the subject should draw the induced pain area on a digital bodychart using the Navigate Pain application (Navigate Pain, Aalborg University, Denmark).

SECONDARY OUTCOMES:
Fibromyalgia Impact Quality-of-Life. | Baseline.
  It will be measured with the version adapted to the Spanish of the Fibromyalgia Impact Questionnaire (FIQ).
Anxiety. | Baseline.
  The version adapted to Spanish from the State Scale (STAI-ES) of the State-Trait Anxiety Inventory (STAI) will be used.
Pain catastrophizing. | Baseline.
  The Spanish version of the Pain Catastrophizing Scale (PCS) will be used.
Depression. | Baseline.
  The adaptation to the Spanish of Beck Depression Inventory II will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain